CLINICAL TRIAL: NCT06813898
Title: ENLIGHTEN: Detection by POSLUMA Following Negative Other PET-PSMA Imaging
Brief Title: An Investigational Scan (rhPSMA-7.3 PET/CT) for Detecting Biochemically Recurrent Prostate Cancer, ENLIGHTEN Trial
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NU 24U08; NCI-2024-09380 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00222061; NU 24U08 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Masking Description: Reads will be completed by three trained radiologists blinded to each other's reads.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (rhPSMA-7.3 PET/CT) (Experimental): Patients receive rhPSMA 7.3 IV and undergo PET/CT 60 minutes later on day 1.
  Interventions: Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Flotufolastat F-18 Gallium; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Other: Flotufolastat F-18 Gallium — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 Radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; Posluma; rhPSMA-7.3 (18F)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial evaluates an imaging technique (rhPSMA-7.3 positron emission tomography [PET]/computed tomography [CT]) for detecting prostate cancer in patients who have increasing prostate-specific antigen levels following prior treatment (biochemical recurrence) but who were prostate specific membrane antigen negative on their most recent PET scan. Contrast agents like rhPSMA-7.3 (also called POSLUMA) circulate in the blood until they find their intended target. Once they are taken up by the target tumor cells, they can be visualized using PET/CT cameras. A PET scan is a procedure in which a small amount of radioactive tracer (in this case rhPSMA-7.3) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the tracer is taken up. Because tumor cells often take up more tracer than normal cells, the pictures can be used to find tumor cells in the body. A CT scan is a procedure that uses a computer linked to an x-ray machine to make a series of detailed pictures of areas inside the body. The pictures are taken from different angles and are used to create 3-dimensional views of tissues and organs. Combining a PET scan with a CT scan can help make the image easier to interpret. PET/CT scans are hybrid scanners that combine both modalities into a single scan during the same examination. The researchers want to determine whether the rhPSMA7.3 PET/CT scan is useful for detecting biochemically recurrent prostate cancer in patients who were negative on prior non-POSLUMA PET imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine consensus detection rate by flotufolastat F-18 gallium (rhPSMA-7.3)-PET (POSLUMA) scan in men with recent negative non-POSLUMA PET prostate specific membrane antigen (PSMA) scans.

SECONDARY OBJECTIVES:

I. Determine patient level verified detection rates (by histopathology or a surrogate standard of truth [second contemporaneous imaging, treatment response/change in subsequent imaging]).

II. Determine change in management plan based on POSLUMA scan (major / minor).

EXPLORATORY OBJECTIVE:

I. Determine patient and patient disease characteristics consistent with a positive POSLUMA scan at prostate specific antigen (PSA) < 0.5ng/ml (i.e. pathological Gleason grade, PSA at scan, time to biochemical recurrence [BCR], prostate-specific antigen doubling time [PSADT]).

OUTLINE:

Patients receive rhPSMA-7.3 intravenously (IV) and undergo PET/CT 60 minutes later on day 1.

After completion of study intervention, patients are followed up at 14 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Men with a history of prostate adenocarcinoma treated with local therapy (including radical prostatectomy or radical prostatectomy and secondary therapy [i.e. salvage radiation])
* Men must have biochemical recurrence (defined as PSA >= 0.1ng/ml) after therapy
* PSA < 0.5ng/ml (within 90 days of enrollment)
* Men must have had negative or equivocal PET PSMA based imaging with 90 days of enrollment with an Food and Drug Administration (FDA) approved non-POSLUMA tracer
* Non-castrate testosterone (testosterone [T] > 50ng/dL) within 90 days of study entry
* Institutional Review Board (IRB)-/Independent Ethics Committee (IEC)-approved written informed consent and privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on the study
* Concurrent diseases and malignancies are permitted

Exclusion Criteria:

* Most recent PSA not between 0.1ng/ml and 0.5ng/ml
* Men with non-metastatic castrate resistant prostate cancer (defined as rising PSA and T < 50ng/dl)
* Patients receiving 5-alpha reductase inhibitors, androgen deprivation therapy and androgen receptor antagonists within 3 months of enrollment (men may start these therapies at physician discretion immediately following POSLUMA PET PSMA scan)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Consensus detection rate | Up to 2 years
  Reads will be completed for the positron emission tomography (PET)/computed tomography (CT) by three trained radiologist blinded to each other's read. Uptake values of rhPSMA-7.3 (POSLUMA) in the prostate bed and other sites (i.e. lymph nodes or bones) will be evaluated. Location and avidity (standardized uptake value) of all identified PET positive sites will be recorded (series/slice number). Consensus read will be determined as positive or negative at the patient level as the consensus of at least 2 of the 3 reading radiologists. Detection rates will be presented with 95% confidence intervals.

SECONDARY OUTCOMES:
Patient level verified detection rates | Up to 2 years
  Patient level verified detection rates will be assessed directly by histopathology or indirectly by secondary imaging or serial imaging with treatment response over the course of 2 years from study scan. Results will be reported in tabular format.
Change in management plan based on POSLUMA scan | Up to 2 years
  The change in management plan based on POSLUMA scan will be assessed as no, minor, or major change as dictated at provider's discretion after POSLUMA scan. Decisions regarding the care of the patient following PET/CT will be made and change from the pre-scan clinical pathway will be recorded subjectively by the treating physician as none, minor or major. Minor changes would include changes in intended frequency of monitoring, modifications within a radiation treatment field. Major changes would include changing from observation to treatment, treatment to observation, extension or inclusion of a new radiation treatment field, extension or reduction in duration of or use of additional systemic medications. Changes in management plans will be reported as frequencies and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Ross, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States